CLINICAL TRIAL: NCT04451980
Title: The HIV, Adipose Tissue Immunology, and Metabolism Study
Acronym: HATIM
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, John R. Koethe, Assistant Professor, Infectious Disease - Medicine, Vanderbilt University Medical Center
Other Study IDs: 161254
Record Dates: First submitted 2020-06-16; First posted 2020-06-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hiv; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collection and retention of whole adipose tissue samples, adipose tissue stromal vascular fraction, peripheral blood mononuclear cells, and plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (4):
- HIV+ non-diabetics: HIV-infected participants with hemoglobin A1c (HbA1c) <5.7% or fasting glucose <100 mg/dl.
  Interventions: Procedure: Subcutaneous adipose tissue biopsy; Radiation: CT scan; Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Blood collection
- HIV+ pre-diabetics: HIV-infected participants with HbA1c 5.7-6.4% or fasting glucose 100-125 mg/dl.
  Interventions: Procedure: Subcutaneous adipose tissue biopsy; Radiation: CT scan; Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Blood collection
- HIV+ diabetics: HIV-infected participants with HbA1c >=6.5% or fasting glucose >=126 mg/dl or on anti-diabetic medications.
  Interventions: Procedure: Subcutaneous adipose tissue biopsy; Radiation: CT scan; Diagnostic Test: Blood collection
- HIV-negative diabetics: HIV-negative participants with HbA1c >=6.5% or fasting glucose >=126 mg/dl or on anti-diabetic medications.
  Interventions: Procedure: Subcutaneous adipose tissue biopsy; Radiation: CT scan; Diagnostic Test: Blood collection

INTERVENTIONS:
Procedure: Subcutaneous adipose tissue biopsy — Percutaneous adipose tissue biopsy
Radiation: CT scan — CT scan of chest and abdomen without contrast
Diagnostic Test: Oral glucose tolerance test — Ingestion of 75g of oral glucose syrup and measurement of blood glucose and insulin at time 0, 15 min, 30 min, 60 min, 90 min, and 120 min.
  Groups: HIV+ non-diabetics; HIV+ pre-diabetics
Diagnostic Test: Blood collection — Fasting blood collection for plasma cytokines and T cell phenotypes.

SUMMARY:
With the introduction of effective anti-retroviral therapy (ART), HIV-infected persons can now survive for decades, but this success has been accompanied by an increased risk of developing metabolic disease and diabetes in HIV-infected persons compared to the general population. Recent studies from HIV-negative subjects have identified several associations between circulating immune cell populations and impaired glucose tolerance, including increased activated CD4+ and CD8+ T cells, and reduced regulatory T cells. Of note, these same changes in peripheral T cell subsets are frequently observed in patients with chronic HIV infection. The goal of this study is to assess whether the circulating T cell distribution is reflective of the adipose tissue T cell distribution, and to understand whether chronic adipose tissue T cell activation may impair adipocyte (i.e., fat cell) function and insulin sensitivity. If the investigators' hypotheses are correct, this will demonstrate that chronic peripheral immune activation (i.e., high memory T cells, low naïve cells, and increased expression of activation surface markers) is associated with greater adipose-resident CD4+ and CD8+ T cell expression of activation markers, adipose tissue inflammation, and insulin resistance.

DETAILED DESCRIPTION:
With the introduction of effective antiretroviral therapy (ART), HIV-infected persons can now survive for decades, but this success has been accompanied by an increased risk of developing metabolic disease compared HIV-negative persons. In the Multicenter AIDS Cohort Study, HIV-infected men had a greater than 4-fold increased incidence of a new diabetes diagnosis compared to HIV-negative men after adjusting for age and body mass index (BMI). Prevalence studies of diabetes in HIV-infected individuals on ART have reported incidence rates of 3.1 to 14 per 1000 patient-years. Furthermore, treated HIV infection appears to act synergistically with other risk factors, and diabetes prevalence is especially high among HIV-infected individuals with high BMI and advanced age.

Recent studies from HIV-negative subjects identified several associations between adaptive immune cell populations and impaired glucose tolerance. Peripheral T regulatory (Treg) cells are significantly lower in patients with type-2 diabetes , while the numbers activated T cells, CD4+ TH1 (pro-inflammatory) cells, and memory CD4+ T cells are higher in diabetics.

Immune cells translocate from the circulation into adipose tissue in a dynamic process, and T cells are present in the stromal fraction of adipose tissue and affect adipocyte function. The striking increase in adipose tissue CD4+ TH1 cells and CD8+ T cells, and a decrease in Treg cells, observed in obesity may have an important role in the development of insulin resistance. Secretion of the proinflammatory cytokines interferon-γ and interleukin (IL)-17 by TH1 and TH17 cells are implicated in the induction of proinflammatory M1 macrophages, which express IL-6 and tumor necrosis factor alpha, and inhibit adipocyte insulin signaling by promoting phosphorylation of insulin receptor substrate 1. The investigators hypothesize that the chronic, HIV-related activation of circulating CD4+ and CD8+ T cells may be accompanied by the accumulation of activated T cells in adipose tissue with adverse effects on metabolic activity.

In this study, the investigators will test the hypothesis that the oligoclonal expansion of chronically activated peripheral T cells in adipose tissue is a primary driver of macrophage inflammation and reduced adipocyte insulin sensitivity. Furthermore, the investigators propose that this represents a central mechanistic linkage underlying the association between circulating T cell activation and incident diabetes risk observed in HIV-infected and HIV-negative individuals.

ELIGIBILITY:
HIV+ Participants:

Inclusion Criteria:

* On antiretroviral therapy for at least 18 months
* HIV-1 RNA <400 copies/ml for the prior 12 months
* CD4+ count >350 cells/µl in the prior 12 months
* HbA1c in prior 6 months within specified limits (See Figure)
* Pre-menopausal by self-report or post-menopausal but not on hormone replacement therapy (HRT)

Exclusion Criteria:

* Known inflammatory or rheumatologic conditions
* Heavy alcohol (>11 drinks per week) or cocaine, amphetamine, or illicit (non-prescribed) opiate abuse by self-report
* Current use of DPP-4 inhibitors.

HIV-negative Participants:

Inclusion Criteria:

* A HbA1c >6.5% or a fasting glucose >126mg/dl, or on anti-diabetic medications for at least 6 months
* Pre-menopausal by self-report or post-menopausal but not on hormone replacement therapy (HRT)

Exclusion criteria:

* Known inflammatory or rheumatologic conditions
* Heavy alcohol (>11 drinks per week) or cocaine, amphetamine, or illicit (non-prescribed) opiate abuse by self-report
* Current use of DPP-4 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-positive participants are recruited from the Vanderbilt Comprehensive Care Clinic, and HIV-negative participants are recruited from Vanderbilt University Medical Center clinics
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue T cell surface marker phenotype and antigen receptor sequence | At study enrollment
  Flow cytometry measurement of adipose tissue T cell surface marker phenotypes and sequencing of T cell receptors, compared by HIV and diabetes status

SECONDARY OUTCOMES:
CT measurements of visceral, hepatic, and pericardial fat content | At study enrollment
  Quantification of visceral, hepatic, and pericardial adipose tissue content, compared by HIV and diabetes status
Circulating T cell surface marker phenotype | At study enrollment
  Flow cytometry measurement of circulating T cell surface marker phenotypes, compared by HIV and diabetes status

CONTACTS AND LOCATIONS:
Overall Officials: John Koethe, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Result] Wanjalla CN, McDonnell WJ, Barnett L, Simmons JD, Furch BD, Lima MC, Woodward BO, Fan R, Fei Y, Baker PG, Ram R, Pilkinton MA, Mashayekhi M, Brown NJ, Mallal SA, Kalams SA, Koethe JR. Adipose Tissue in Persons With HIV Is Enriched for CD4+ T Effector Memory and T Effector Memory RA+ Cells, Which Show Higher CD69 Expression and CD57, CX3CR1, GPR56 Co-expression With Increasing Glucose Intolerance. Front Immunol. 2019 Mar 19;10:408. doi: 10.3389/fimmu.2019.00408. eCollection 2019. PMID 30941121
- [Result] Koethe JR, McDonnell W, Kennedy A, Abana CO, Pilkinton M, Setliff I, Georgiev I, Barnett L, Hager CC, Smith R, Kalams SA, Hasty A, Mallal S. Adipose Tissue is Enriched for Activated and Late-Differentiated CD8+ T Cells and Shows Distinct CD8+ Receptor Usage, Compared With Blood in HIV-Infected Persons. J Acquir Immune Defic Syndr. 2018 Feb 1;77(2):e14-e21. doi: 10.1097/QAI.0000000000001573. PMID 29040163
- [Derived] Bailin SS, Ma S, Perry AS, Terry JG, Carr JJ, Nair S, Silver HJ, Shi M, Mashayekhi M, Kropski JA, Ferguson JF, Wanjalla CN, Das SR, Shah R, Koethe JR, Gabriel CL. The Primacy of Adipose Tissue Gene Expression and Plasma Lipidome in Cardiometabolic Disease in Persons With HIV. J Infect Dis. 2025 Feb 20;231(2):e407-e418. doi: 10.1093/infdis/jiae532. PMID 39657693
- [Derived] Swartz AZ, Robles ME, Park S, Esfandiari H, Bradshaw M, Koethe JR, Silver HJ. Cardiometabolic Characteristics of Obesity Phenotypes in Persons With HIV. Open Forum Infect Dis. 2024 Jul 8;11(7):ofae376. doi: 10.1093/ofid/ofae376. eCollection 2024 Jul. PMID 39035569
- [Derived] Werede AT, Terry JG, Nair S, Temu TM, Shepherd BE, Bailin SS, Mashayekhi M, Gabriel CL, Lima M, Woodward BO, Hannah L, Mallal SA, Beckman JA, Li JZ, Fajnzylber J, Harrison DG, Carr JJ, Koethe JR, Wanjalla CN. Mean Coronary Cross-Sectional Area as a Measure of Arterial Remodeling Using Noncontrast CT Imaging in Persons With HIV. J Am Heart Assoc. 2022 Dec 6;11(23):e025768. doi: 10.1161/JAHA.122.025768. Epub 2022 Nov 16. PMID 36382956

DOCUMENTS (1):
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04451980/Prot_000.pdf